CLINICAL TRIAL: NCT07398586
Title: The Association Between Interleukin-7 Receptor Gene Polymorphism and the Risk of Ulcerative Colitis as Well as the Response to Vedolizumab
Brief Title: The Association Between Interleukin-7 Receptor Gene Polymorphism and the Risk of Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2025-01-130
Record Dates: First submitted 2026-01-05; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis (UC)
Keywords: colitis; ulcerative
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Ulcer | interventions — vedolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC patients (Experimental): Some UC patients received intravenous injection of VDZ (300mg/time) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of VDZ every 8 weeks to maintain treatment.
  Interventions: Biological: Vedolizumab
- normal control (No Intervention): no biological agents treatment

INTERVENTIONS:
Biological: Vedolizumab — Intravenous injection of VDZ (300mg/time) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of VDZ every 8 weeks to maintain treatment.
  Arms: UC patients

SUMMARY:
From January 2020 to December 2024, diagnosed ulcerative colitis(UC) patients and gender- and age-matched normal controls were enrolled from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Investigators' aim is to investigate the associations of IL-7R gene polymorphisms with the risk and clinicopathological characteristics of UC, and to analyze the effects of IL-7R gene variations on the clinical response of vedolizumab(VDZ) treatment in UC patients.

DETAILED DESCRIPTION:
From January 2020 to December 2024, diagnosed UC patients and gender- and age-matched normal controls were enrolled from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Genotypes of IL-7R were determined by multiplex polymerase chain reaction-ligase detection reaction technique. Chi-square test and unconditional logistic regression model were used to analyze the difference in distribution of IL-7R gene polymorphisms between UC group and normal control group, as well as the effects of IL-7R gene variations on the clinicopathological characteristics and 14-week clinical response to VDZ treatment of participants.

ELIGIBILITY:
Inclusion Criteria:

-diagnosed UC based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

-rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 898 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Genotypes of IL-7R | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No